CLINICAL TRIAL: NCT07113600
Title: A Randomized Comparative Study Between Ultrasound Guided Erector Spinae Plane Block and Ultrasound Guided Iliohypogastric/ Ilioinguinal Nerve Block for Postoperative Pain Relief in Female Patients Undergoing Open Hysterectomy
Brief Title: Erector Spinae Plane Block Versus Iliohypogastric/Ilioinguinal Nerve Block for Post-Hysterctomy Pain Relief
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mai Ahmed Ali Mohamed El-sayed, Assistant Professor Of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-119_2023/MSc
Record Dates: First submitted 2025-07-22; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain, Acute
Keywords: Humans; Female; Anesthesia, Conduction; Ultrasonography; Nerve Block; Pain, Postoperative; Ultrasonography, Interventional
MeSH Terms: conditions — Pain, Postoperative | interventions — Nerve Block

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated with a 1:1 allocation ratio into two groups in a parallel manner:
  * Group A(n=29): Patients will receive bilateral ESP block using 20 ml bupivacaine 0.25% on each side.
  * Group B(n=29): Patients will receive bilateral Iliohypogastric and Ilioinguinal nerve block using 20 ml bupivacaine 0.25% on each side.
Who Masked: Participant
Masking Description: Both blocks will be performed after induction of general anesthesia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB (Active Comparator): Patients will receive bilateral Erector Spinae Plane block using 20ml bupivacaine 0.25% on each side.
  Interventions: Other: Nerve Block
- Ilioinguinal/iliohypogastric (Active Comparator): Patients will receive bilateral Iliohypogastric and Ilioinguinal nerve block using 20ml bupivacaine 0.25% on each side.
  Interventions: Other: Nerve Block

INTERVENTIONS:
Other: Nerve Block — Ilioinguinal/ Iliohypogastric nerve block:
  In the supine position, the ultrasound probe probe is positioned in a transverse manner, superior to the anterior superior iliac spine. The three anterior abdominal muscle layers are identified, and the two nerves are identified in the abdominal neurovascular plane.
  A echogenicneedle is inserted in a medial-to-lateral direction. After negative aspiration, 5 ml saline is injected to ensure correct needle tip position then 20 ml of bupivacaine 0.25% is injected gradually close to the nerves.
  Erector spinae plane block:
  In a lateral position, the erector spinae is visualized about 3 cm lateral to T7-T9 spinous processes on the target side. A echogenic needle (50 mm/22 gauge) is advanced in a cephalad to caudad direction until the tip reaches the plane deep to the erector spinae muscle immediately lateral to the transverse process. A 20 ml bupivacaine 0.25% is injected gradually into this plane.

SUMMARY:
The goal of this clinical trial is to compare the degree of pain relief between two techniques of regional anesthesia given to ladies undergoing hysterectomy under general anesthesia.

One group of patients will have a local anesthetic injected between muscle layers in their back (ultrasound guided Erector Spinae plane Block).

The other group will have a local anesthetic injected around specific nerves in their abdomen (ultrasound guided Ilio-hypogastric / ilio-inguinal nerve block ).

Researchers will compare the duration of postoperative pain relief , the degree of pain relief and any possible side effects of either techniques.

DETAILED DESCRIPTION:
The use of ultrasound for the placement of peripheral nerve blocks has received a great deal of attention in anesthesiology literature as well as clinical practice. Advantages of ultrasound-guided regional anesthesia include easy learning, fast onset, higher success rates, more complete blocks, using lower local anesthetic volumes and more safety. Good postoperative analgesia can prevent morbidity associated with abdominal hysterectomy by allowing pain-free, early ambulation and decreasing the risks of long hospital stay such as thrombo-embolism, and other poor outcomes. Truncal blocks such as transversus abdominis plane (TAP) blocks have seen limited success due to shorter duration and sub-optimal analgesia. The ultrasound (US)-guided erector spinae plane block (ESPB) w gained wide attention as a fast procedure that carries a lower risk of hypotension, can be used in patients with coagulopathy, is easy to perform, and requires less training. It provides extensive, potent unilateral analgesia, is performed by local anesthetic injection in the plane between the erector spinae muscle and the Transverse process of the corresponding vertebra. The local anesthetic diffuses into the para vertebral space through spaces between adjacent vertebrae and blocks both the dorsal and ventral branches of the thoracic spinal nerves. Bilateral ESPB performed at low thoracic levels was recently shown to provide satisfactory analgesia for gynecologic and abdominal surgery.

Abdominal field blocks, such as the ilio-inguinal / ilio-hypogastric (IL-IH) nerve block are well- known as simple ways to give long-lasting pain relief and limit narcotic usage after surgery.

The ilio-inguinal and ilio-hypogastric nerves are T 12 and L 1 branches that supply the inguinal region and run between the internal oblique and transversus abdominis muscles, slightly above the anterior superior iliac spine.

The aim of this study is to compare the analgesic effect of ilio-hypogastric / ilio-inguinal versus erector spine plane block on female patients undergoing open hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients above the age of 35 years.
* American Society of Anesthesiologists (ASA) physical status I-II.

Exclusion Criteria:

* Patient refusal.
* History of allergy or intolerance to study medications.
* Chronic opioid use (>3 months).
* Severe renal or hepatic impairment.
* Patients with coagulopathy disorders.
* Infection at injection sites.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The time to first call for analgesia. | The first 12 postoperative hours
  The period of time starting from extubation until the patient asks for analgesia in hours.

SECONDARY OUTCOMES:
postoperative pain score | VAS was assessed at 0, 2, 6, and 12 hours postoperatively.
  Visual analog scale (0-100 mm)
intraoperative hemodynamic changes | Operative time
  Increase in heart rate(beat/min) or systolic blood pressure(mmHg) more than 20% of the baseline , hypotension (defined as a decrease in mean arterial pressure > 25% from the baseline value or systolic arterial pressure < 100 mmHg),

OTHER OUTCOMES:
Total post-operative opioid consumption | The first 12 postoperative hours
  The total Rescue analgesia boluses of morphine ( 0.1mg/kg if the VAS exceeded 3 & repeated until the VAS dropped below 3.